CLINICAL TRIAL: NCT02995330
Title: A Pilot Study of Sex-Mismatched Allogeneic Bone Marrow Transplantation for Men With Metastatic Castration-Resistant Prostate Cancer
Brief Title: Sex-Mismatched Allogeneic Bone Marrow Transplantation for Men With Metastatic Castration-Resistant Prostate Cancer
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: lack of accrual
Sponsor: Sidney Kimmel Comprehensive Cancer Center at Johns Hopkins (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: J1608; IRB00086105 (Other: JHMI-IRB)
Record Dates: First submitted 2016-12-14; First posted 2016-12-16 (Estimated); Results first posted 2024-02-13 (Actual); Last update posted 2024-02-13 (Actual); Status verified 2024-02

CONDITIONS: Prostate Cancer
Keywords: Metastatic Castration-Resistant Prostate Cancer; Bone Marrow Transplantation
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Bone Marrow Transplantation; Cyclophosphamide; testosterone 17 beta-cypionate; Testosterone

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Bone marrow transplantation (Experimental): Bone marrow transplantation followed by Cytoxan and testosterone
  Day -6 to -1: Subjects will be treated with a standard non-myeloablative conditioning regimen
  Day 0: subjects will be infused with non-T-cell depleted bone marrow from a related female donor.
  Subjects will receive GVHD prophylaxis consisting of:
  Day +3 and +4: Cytoxan (Cy) 50mg/kg IV Day +5 through Day +180: tacrolimus (IV or PO) beginning [dose adjusted to maintain trough level of 5-15 ng/mL] Day +5 through Day +35: Mycophenolate mofetil (MMF) 15 mg/kg PO TID, with a maximum dose of 1g TID.
  Day +5: filgrastim (G-CSF) 5 mcg/kg/day, continued until ANC ≥ 1500/mm3.
  Day +60, +90, and +120: testosterone cypionate 400 mg IM every 30 days x 3 doses
  Subjects will be maintained on continuous LHRH agonist/antagonist therapy (if not previously surgically castrated). Subjects who achieve biochemical CR will stop LHRH agonist/antagonist treatmentat day 180.
  Interventions: Procedure: Bone marrow transplantation; Drug: Cytoxan; Drug: testosterone cypionate

INTERVENTIONS:
Procedure: Bone marrow transplantation — Infused with non-T-cell depleted bone marrow from a related female donor on Day 0
Drug: Cytoxan — Cytoxan 50mg/kg IV on Days +3 and +4
Drug: testosterone cypionate — testosterone cypionate 400 mg IM will be administered on Day +60, +90, and +120 (every 30 days x 3 doses)
  Other Names: testosterone

SUMMARY:
Men with progressive metastatic Castration-Resistant Prostate Cancer post first-line treatment with either androgen deprivation therapy alone or androgen deprivation therapy plus docetaxel who have an identified related female donor (mother sister, daughter, second degree relative such as granddaughter or niece) will undergo bone marrow transplantation followed by post-transplant Cytoxan (PT/Cy) and testosterone.

DETAILED DESCRIPTION:
Men will undergo pre-transplant screening evaluation and be enrolled in the study. Subjects will be treated with a standard non-myeloablative conditioning regimen consisting of Fludarabine 30 mg/m2 IV Days -6 to -2; Cy 14.5 mg/kg IV Days -6 and -5; Total body irradiation (TBI) 200 cGy Day -1. On Day 0, patients will be infused with non-T-cell depleted bone marrow from a related female donor. Patients will receive GVHD prophylaxis consisting of: Cy 50mg/kg IV on Days +3 and +4; tacrolimus (IV or PO) beginning on Day +5 [dose adjusted to maintain trough level of 5-15 ng/mL] through day+180; Mycophenolate mofetil (MMF) 15 mg/kg PO TID, with a maximum dose of 1g TID beginning on Day +5 through Day +35. Patients will receive filgrastim (G-CSF) 5 mcg/kg/day beginning on Day +5 and continued until ANC ≥ 1500/mm3. Lastly, to produce maintenance tumor antigen stimulation, patients will be maintained on continuous LHRH agonist/antagonist therapy (if not previously surgically castrated) to suppress endogenous testosterone production throughout the treatment period; testosterone cypionate 400 mg IM will be administered on Day +60, +90, and +120 (every 30 days x 3 doses). Patients who achieve biochemical CR will stop LHRH agonist/antagonist treatment at day 180. Patients will be followed for 3 years post-BMT.

ELIGIBILITY:
Inclusion Criteria:

* Performance status ≤1
* Age ≥18 years and ≤ 75 years old
* Histologically-confirmed adenocarcinoma of the prostate
* Treated with continuous androgen ablative therapy (either surgical castration or LHRH agonist/antagonist) with documented castrate level of serum testosterone (<50 ng/dl)
* Metastatic disease radiographically documented by CT or bone scan
* Patient must be HLA typed at high resolution using DNA based typing at the following loci: HLA-A, -B, -C, and DRB1
* Patient must have available one or more potential first (biologic mother, sister, half-sister, or daughter) or second-degree related female donor. Mothers and daughters have a 100% chance of being haploidentical matches, sisters a 75% chance of being matched or haploidentical, and second degree relatives have a 50% chance of being haploidentical matches. The donor and recipient must be HLA identical for at least one antigen at HLA-A, -B, -C and HLA-DRB1.
* Screening PSA must be ≥ 1.0 ng/mL.
* Prior therapy with one second line hormonal therapy is allowed (i.e. bicalutamide, nilutamide, flutamide, ketoconazole, abiraterone, enzalutamide, ARN-509).
* Prior docetaxel (≤ 6 cycles) as first line therapy
* Cardiac ejection fraction at rest must be ≥ 40%
* Acceptable liver function: Bilirubin < 2.5 mg/dL (unless due to Gilbert's disease, AST (SGOT) and ALT (SGPT) < 5 times upper limit of normal.
* Acceptable renal function: Serum creatinine within normal range.
* Pulmonary function: DLCO (corrected for hemoglobin), FEV1 and FVC >50% predicted.
* At least 4 wks since prior radiation or surgery with full recovery (no persistent toxicity ≥ Grade 1)
* Ability to understand and willingness to sign a written informed consent document.

Exclusion Criteria:

* Prior treatment with Sipuleucel-T, radium-223, strontium-89, or samarium-153
* Prior chemotherapy (docetaxel, cabazitaxel) for castrate resistant prostate cancer
* Evidence of serious and/or unstable pre-existing medical, psychiatric or other condition (including laboratory abnormalities) that could interfere with patient safety or provision of informed consent to participate in this study
* Active uncontrolled infection, including known history of HIV/AIDS or hepatitis B or C.
* Any psychological, familial, sociological, or geographical condition that could potentially interfere with compliance with the study protocol and follow-up schedule.

Ages: 18 Years to 75 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3 (Actual)
Dates: Start 2017-02-09 (Actual); Primary Completion 2021-06-16 (Actual); Study Completion 2021-06-16 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Samuel Denmeade, MD, Principal Investigator — Johns Hopkins University
Locations (1):
- Johns Hopkins Hospital, Baltimore, Maryland, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Bone Marrow Transplantation: Bone marrow transplantation followed by Cytoxan and testosterone
  Day -6 to -1: Subjects will be treated with a standard non-myeloablative conditioning regimen
  Day 0: subjects will be infused with non-T-cell depleted bone marrow from a related female donor.
  Subjects will receive GVHD prophylaxis consisting of:
  Day +3 and +4: Cytoxan (Cy) 50mg/kg IV Day +5 through Day +180: tacrolimus (IV or PO) beginning [dose adjusted to maintain trough level of 5-15 ng/mL] Day +5 through Day +35: Mycophenolate mofetil (MMF) 15 mg/kg PO TID, with a maximum dose of 1g TID.
  Day +5: filgrastim (G-CSF) 5 mcg/kg/day, continued until ANC ≥ 1500/mm3.
  Day +60, +90, and +120: testosterone cypionate 400 mg IM every 30 days x 3 doses
  Subjects will be maintained on continuous LHRH agonist/antagonist therapy (if not previously surgically castrated). Subjects who achieve biochemical CR will stop LHRH agonist/antagonist treatmentat day 180.
  Bone marrow transplantation: Infused with non-T-cell depleted bone marrow from a related female donor on Day 0
  Cytoxan: Cytoxan 50mg/kg IV on Days +3 and +4
  testosterone cypionate: testosterone cypionate 400 mg IM will be administered on Day +60, +90, and +120 (every 30 days x 3 doses)
Period: Overall Study
Arm/Group | Bone Marrow Transplantation
Started | 3
Completed | 3
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Bone Marrow Transplantation
Number analyzed (Participants) | 3
Age, Continuous [Mean (Full Range); unit: years] | 58 [48 to 64]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 3
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 1
  White | 2
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 3

OUTCOME MEASURES:

1. Primary Outcome: Prostate-specific Antigen (PSA) Response
Description: Percentage of participants with complete biochemical response at 6 months post-transplant (prostate-specific antigen <0.1 ng/mL for patients post-prostatectomy and prostate-specific antigen< 1 ng/mL for patients post-radiation therapy)
Time Frame: 6 months
Measure: Number; unit: percent of participants
Arm/Group | Bone Marrow Transplantation
Number analyzed (Participants) | 3
percent of participants | 0

2. Secondary Outcome: Transplant-related Mortality
Description: Number of participants who experience transplant-related mortality (TRM) following alloBMT
Time Frame: 3 years
Measure: Number; unit: participants
Arm/Group | Bone Marrow Transplantation
Number analyzed (Participants) | 3
participants | 0

3. Secondary Outcome: Number of Participants With a Prostate-specific Antigen Decline ≥ 50%
Description: Proportion of patients achieving a prostate-specific antigen decline ≥ 50% according to Prostate Cancer Working Group (PCWG2) criteria
Time Frame: 3 years
Measure: Count of Participants; unit: Participants
Arm/Group | Bone Marrow Transplantation
Number analyzed (Participants) | 3
Participants | 1

4. Secondary Outcome: Objective Response Rate or Either Complete Response (CR) or Partial Response (PR)
Description: Percentage of participants with reduction in measurable disease on CT scan as defined by RECIST criteria: Complete Response (CR)= disappearance of all target lesions; Partial Response (PR)= at least a 30% decrease in the sum of the largest diameter (LD) of target lesions, taking as reference the baseline sum LD; Progressive Disease (PD)= at least 20% increase in the sum of the LD of target lesions, taking as reference the smallest sum LD recorded since the treatment started or the appearance of one or more new lesions; Stable disease (SD)= Neither sufficient shrinkage to qualify for PR nor sufficient increase to qualify for PD, taking as reference the smallest sum LD since the treatment started
Time Frame: 3 years
Measure: Count of Participants; unit: Participants
Arm/Group | Bone Marrow Transplantation
Number analyzed (Participants) | 3
Participants | 0

5. Secondary Outcome: Time to PSA Progression
Description: Time to PSA progression as defined by PCWG2 criteria ( PSA progression as an increase in PSA greater than 25% and >2 ng/ml above nadir, confirmed by progression at 2 timepoints at least 3 weeks apart)
Time Frame: 3 years
Population: This data was not collected because the study closed before the time to PSA progression could be assessed
Arm/Group | Bone Marrow Transplantation
Number analyzed (Participants) | 0

6. Secondary Outcome: Time to Clinical/Radiographic Progression
Description: Time to clinical/radiographic progression on CT and bone scan as defined by RECIST ( >=25% increase in PSA from nadir (and by >=2ng/mL), and/or clinical/radiographic progression (clinical progression = symptomatic progression, worsening of disease-related symptoms or new cancer-related complications; radiographic progression on CT scan defined by RECIST 1.1 criteria: >=20% enlargement in sum diameter of soft-tissue target lesions; or on bone scan >=1 new bone lesions), initiation of ADT or death due to any cause, whichever occurs first.) and PCWG2 criteria ( PSA progression as an increase in PSA greater than 25% and >2 ng/ml above nadir, confirmed by progression at 2 timepoints at least 3 weeks apart), respectively.
Time Frame: 3 years
Population: This data was not collected because the study closed before the time to Clinical/radiographic progression could be assessed
Arm/Group | Bone Marrow Transplantation
Number analyzed (Participants) | 0

7. Secondary Outcome: Number of Participants Who Experience Acute Graft-versus-host-disease (GVHD)
Description: Number of participants with acute GVHD grades 2-4 and grades 3-4 as defined by Przepiorka criteria. Przepiorka criteria stages the degree of organ involvement in the skin, liver and gastrointestinal (GI) tract, based on severity, with Stage 1+ being least sever and Stage 4+ being most severe. Grading of acute GVHD is as follows: Grade I (skin involvement stages 1+ to 2+, with no liver or GI involvement), Grade II (skin involvement stages 1+ to 3+, liver 1+, GI tract 1+), Grade III (skin involvement stages 2+ to 3+, liver 1+, GI tract 2+ to 4+), Grade IV (skin involvement stages 4+, liver 4+)
Time Frame: 3 years
Measure: Count of Participants; unit: Participants
Arm/Group | Bone Marrow Transplantation
Number analyzed (Participants) | 3
Participants | 2

8. Secondary Outcome: Number of Participants Who Experience Chronic GVHD
Description: Number of participants who experience chronic GVHD (defined as cGVHD progression while on prednisone at ≥1 mg/kg/day for 1-2 weeks, or stable cGVHD while on ≥0.5 mg/kg/day for 1-2 months, and additional patients remain steroid-dependent with repeated symptom flares during taper of corticosteroids below 0.25 mg/kg/day ) as defined by the protocol.
Time Frame: 3 years
Measure: Count of Participants; unit: Participants
Arm/Group | Bone Marrow Transplantation
Number analyzed (Participants) | 3
Participants | 1

9. Secondary Outcome: Number of Participants With Donor Chimerism
Description: Patients with any amount of donor chimerism around day 60 will be considered as having engrafted. Chimerism determinations will be made on peripheral blood by a number of different methods depending on the specific patient. Methods may include (i) the usual standard of restriction fragment length polymorphism (RFLP) if the donor and recipient RFLPs are informative, (ii) fluorescence in-situ hybridization (FISH) for Y-chromosome markers on PBMC if the donor is male, (iii) cytogenetic analysis, (iv) flow cytometric analysis of HLA-A, B or DR on lymphocytes in the peripheral blood if haploidentical and suitable reagents exist or (v) PCR analysis of variable nucleotide tandem repeats (VNTR) in PBMC if informative. Mixed donor chimerism will be defined as >0%, but <95%. Complete donor chimerism will be defined as >95%. Patients who have relapsed or died prior to day 60 will not be evaluable for full donor chimerism, as these are competing risk factors.
Time Frame: up to 60 days
Measure: Count of Participants; unit: Participants
Arm/Group | Bone Marrow Transplantation
Number analyzed (Participants) | 3
Participants | 3

10. Secondary Outcome: Number of Participants With Graft Failure
Description: Number of participants with failure to engraft due to rejection by host lymphocytes.
Time Frame: 3 years
Measure: Count of Participants; unit: Participants
Arm/Group | Bone Marrow Transplantation
Number analyzed (Participants) | 3
Participants | 0

11. Secondary Outcome: Effects of Post-transplantation Cyclophosphamide on the Immune Reconstitution of T Cells, B Cells, and NK Cells
Description: The number of participants that have a changed to post-transplantation cyclophosphamide on the immune reconstitution of T cells, B cells, and NK cells
Time Frame: 5 years
Population: Samples were collected but the tests were not run due to study closure.
Arm/Group | Bone Marrow Transplantation
Number analyzed (Participants) | 0

12. Secondary Outcome: Number of Participants Who Develop HLA Specific Antibodies
Description: Number of participants who develop HLA specific antibodies after HLA mismatched, allogeneic partially HLA-mismatched bone marrow transplantation
Time Frame: 5 years
Population: Samples were collected but the tests were not run due to study closure.
Arm/Group | Bone Marrow Transplantation
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Time Frame: All Adverse events were only collected for the first 6 months. Then for the next 3 year of follow up only transplant-related mortality (TRM) following alloBMT where collected.
Description: There were no serious adverse events for this study
Arm/Group | Bone Marrow Transplantation
All-Cause Mortality (participants affected / at risk) | 0/3
Serious Adverse Events (participants affected / at risk) | 0/3
Other Adverse Events (participants affected / at risk) | 0/3

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-07-02): https://cdn.clinicaltrials.gov/large-docs/30/NCT02995330/Prot_SAP_000.pdf